CLINICAL TRIAL: NCT01268865
Title: Clinical Application of Acoustic Radiation Force Impulse (ARFI)Technology in Prediction of Liver Fibrosis in HBV and HCV-infected Patients
Brief Title: Acoustic Radiation Force Impulse (ARFI)Technology in Prediction of Liver Fibrosis
Acronym: ARFI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sheng-Hung Chen, China Medical University Hospital
Other Study IDs: DMR99-IRB-240
Record Dates: First submitted 2010-12-30; First posted 2010-12-31 (Estimated); Last update posted 2011-06-03 (Estimated); Status verified 2011-06

CONDITIONS: Liver Fibrosis
Keywords: Acoustic Radiation Force Impulse (ARFI); Virtual Touch Quantification (VTQ); liver stiffness measurement (LSM); liver fibrosis; cirrhosis; hepatitis B; hepatitis C
MeSH Terms: conditions — Liver Cirrhosis; Fibrosis; Hepatitis B; Hepatitis C

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- HBV-infected
- HCV-infected

SUMMARY:
Background: In patients with chronic liver diseases, liver fibrosis staging is crucial for hazard evaluation of future disease complication development and thus for the optimal decision making on treatment selections.In the era of antiviral and antifibrotic treatments, clinical and research demands are also increasing for non-invasive surveillance of liver fibrosis to evaluate the progression or regression. However, local baseline data on liver stiffness measurement (LSM) using ARFI technique is still lacking in Taiwan, where viral hepatitides are highly endemic. Aim: Using the ARFI elastosonography, we are dedicated to the aims to recruit patients based on strict but appropriate criteria, to complete the correlation and validity studies between ARFI quantification and the referenced METAVIR fibrosis scoring and to conduct subsequent innovative studies on liver diseases. Materials and Methods: We plan to perform the ARFI quantification for each HBV or HCV-infected patient immediately followed by priorly scheduled conventional liver biopsy for METAVIR scoring during the same session of examination. Statistics: The first year's study using ARFI will focus on the correlation testings and validity studies using receiver operating characteristics.

DETAILED DESCRIPTION:
Contribution and Future Works: Using the ARFI quantification either as a causal factor or as a outcome, we can conduct future analyses ranging from validations, regressions to prospective time-to-event analysis among our cohorts.

ELIGIBILITY:
Inclusion Criteria:

* infected with HBV only or HCV only

Exclusion Criteria:

* concurrent HBV-HCV infection, etc.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: HBV or HCV-infected patients about to undergo liver biopsy to assist in clinical decision making
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2010-12

CONTACTS AND LOCATIONS:
Overall Officials: Sheng-Hung Chen, MD, Principal Investigator — Hepatogastroenterology, Department of Internal Medicine, China Medical University Hospital; Cheng-Yuan Peng, MD, PhD, Study Director — Hepatogastroenterology, Department of Internal Medicine, China Medical University Hospital
Locations (1):
- China Medical University Hospital, Taichung, Taiwan